CLINICAL TRIAL: NCT01876875
Title: Energy-restricted, n-3 Polysaturated Fatty Acids-rich Diet Improves the Clinical Response to Immuno-modulating Drugs in Obese Patients With Plaque-type Psoriasis: a Randomized Control Clinical Trial.
Brief Title: n-3 Polysaturated Fatty Acids-rich Diet in Psoriasis
Acronym: PSO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Eleonora Riccio, md, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cataldi13; CAT (Other: ethic commettee)
Record Dates: First submitted 2013-06-05; First posted 2013-06-13 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2008-10

CONDITIONS: Plaque-type Psoriasis; Obesity (Body Mass Index >30 kg/m2)
Keywords: psoriasis; obesity
MeSH Terms: conditions — Obesity; Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): The patients of this group were randomized to receive an energy-restricted diet (20 kcal/kg/ideal body weight/day) enriched of n-3 PUFAs (average 2.6 g/d).
  Interventions: Dietary Supplement: Energy-restricted, n-3 polysaturated fatty acids-rich diet
- Control group (Active Comparator): The participants of this group are randomized to receive drug therapy alone, continuing their usual diet
  Interventions: Dietary Supplement: Usual diet

INTERVENTIONS:
Dietary Supplement: Energy-restricted, n-3 polysaturated fatty acids-rich diet — The active diet aimed to reduce body weight, to enhance the total intake of n-3 PUFA and to decrease the total intake of n-6 PUFAs. The diet plan was designed to supply an energy intake of 20 kcal/kg/day to maintain an ideal body weight, and followed the guidelines of the American Heart Association (AHA) 'Step-One' Diet: Carbohydrates (mainly complex carbohydrates) and protein constituted of 50-60% and 10-20% of total calories, respectively, and total fat did not exceed 30% of calories. Food values for energy and nutrients were taken from the tables of the Italian National Institute of Nutrition, Souci's Food Composition and Nutrition Tables and the European Institute of Oncology. For long-term and practical daily eating habits, it was important to easily incorporate and consume a variety of selected foods.
  Arms: Intervention group
Dietary Supplement: Usual diet — The patients of this group were randomized to continue their usual diet
  Arms: Control group

SUMMARY:
Low-grade systemic inflammation associated with obesity may worsen the clinical course of psoriasis. Both a low-calorie diet and nutritional supplementation have been shown to have an impact on the clinical course of psoriasis, including an anti-inflammatory effect of n-3 polyunsaturated fatty acids (PUFAs). This study aimed to assess the effectiveness of an energy-restricted diet, enriched in n-3 PUFAs and poor in n-6 PUFAs, on metabolic markers and clinical outcome of obese patients with psoriasis.

Methods: Forty-four obese patients with mild-to-severe plaque-type psoriasis treated with immuno-suppressive drugs were randomized to assume either their usual diet or an energy-restricted diet (20 kcal/kg/ideal body weight/day) enriched of n-3 PUFAs (average 2.6 g/d). All patients continued their immuno-modulating therapy throughout the study. End-point measures included anthropometric, biochemical and clinical parameters at baseline, 3 and 6 months.

DETAILED DESCRIPTION:
Psoriasis is one of the most common chronic inflammatory skin disorders, affecting about 2% of the general population. It is considered to be a T-cell-mediated inflammatory skin disease which is characterized by hyper-proliferation and poor differentiation of epidermal keratinocytes. Even if the susceptibility to psoriasis is inherited, the inflammatory reaction is modulated by diet, lifestyle and environmental factors such as infections and stress. Polyunsaturated fatty acids (PUFAs) are showing promise as safe adjunctive treatments for many skin disorders, including psoriasis.

There are two main families of PUFAs: n-3 and n-6 PUFAs. Alpha-linolenic acid (ALA) is the only essential n-3 PUFA, while linoleic acid is the only essential n-6 PUFA. These fatty acids form the building blocks for downstream long-chain fatty acids: On the n-6 side, linoleic acid converts to gamma-linolenic acid (GLA) and dihomo-gamma-linolenic acid (DGLA), the latter of which may be converted to either pro-inflammatory arachidonic acid (AA) or anti-inflammatory prostaglandins, prostaglandin E1 (PGE1). AA (which can also be derived from the diet) is primarily a precursor to pro-inflammatory eicosanoids, prostaglandin E2 (PGE2), and leukotrienes and, to a much smaller extent, anti-inflammatory prostacyclin. On the n-3 side, a small amount of ALA converts to eicosapentaenoic acid (EPA), and then to docosahexaenoic acid (DHA). EPA serves primarily as a precursor to anti-inflammatory prostaglandins, prostaglandin E3 (PGE3) and inhibits both the production of AA from DGLA and the production of PGE2 or thromboxane from AA. Skin cells produce eicosanoids in response to various stimuli contributing to inflammatory conditions.The active involvement of fatty acids in skin health and epidermal barrier function justifies the choice of systemic supplementation with n-3PUFA as an effective strategy for the improvement of inflammatory conditions. Epidemiological observations of a lower incidence of autoimmune and inflammatory disorders, including psoriasis, in a population of Greenland Eskimos compared with gender- and age-matched groups living in Denmark provided early suggestive evidence of the important role of n-3 PUFAs dietary intake on inflammation. An improvement in psoriasis has also been observed during daily dietary supplementation with fish oil containing n-3 PUFAs. As mentioned, AA is a pro-inflammatory fatty acid. As a result, a low dietary intake of AA, typical of low-protein and vegetarian diets, may produce a less anti-inflammatory effects. The Western diet is "deficient" in n-3 PUFAs, with an n-6/n-3 ratio of 15/1 to 16/1, as compared to the 1/1 ratio as found in wild animals and presumably human beings prior to the industrial revolution. Although the ability of a low-protein diet to improve symptoms in psoriasis patients has not been consistently supported a remarkable treatment efficacy was reported for a patient by Schamberg. In a case-control study, Naldi et al showed that an increased intake of fresh fruits and certain vegetables was linked to a decreased prevalence of psoriasis, although the mechanism was not clear.

Calorie restriction and/or weight loss may also influence symptom severity in psoriasis. In obese patients with moderate-to-severe plaque psoriasis, weight loss was shown to improve the therapeutic response to cyclosporine. In mice, four weeks of calorie restriction (by 33% of energy intake) led to a decrease of 45% in the epidermal cell proliferation rate. Likewise, symptoms of inflammatory diseases such as rheumatoid arthritis have been shown to be improved through fasting or low-energy diets. Associations have also been recognized between psoriasis and an increased incidence of metabolic syndrome (visceral obesity, diabetes or insulin resistance, hypertension, and dyslipidemia). Although the link between psoriasis and individual components of metabolic syndrome is not completely elucidated, visceral fat, which releases pro-inflammatory cytokines, appears to play a role in both metabolic syndrome and psoriasis.

Additional factors influencing the severity of psoriasis have been examined, such as alcohol consumption. Alcohol may enhance the production of inflammatory cytokines and cell cycle activators, which could lead to epidermal hyperproliferation. Although there is no generally recognized decisive cure for psoriasis, many treatments are commonly used to reduce the severity of symptoms and lessen their impact on the patient's quality of life. For moderate-to-severe psoriasis, phototherapy and topical and/or systemic therapies are the standard medical therapies. Examples include corticosteroids, emollients, tar, methotrexate, and cyclosporine. However, many of these treatments are associated with significant adverse effects. Some alternative systemic therapies include monoclonal antibodies, fumaric acid esters, vitamin D analogs, novel retinoids, macrolactams, and biologic immune modifiers such as anti-tumor necrosis factor (TNF) agents.

The present study explores the effectiveness of an energy-restricted n-3 fatty acid-rich diet on the nutritional and clinical outcome of obese patients with mild-to-severe psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) >30 kg/m2,
* age ≥18 years
* clinical diagnosis of plaque-type psoriasis,
* mild-to-severe psoriasis clinically stable for at least 5 months
* no change in psoriasis therapies for at least five months

Exclusion Criteria:

* diabetes,
* malignancy,
* history of food intolerance or autoimmune disorders,
* patients non-collaborative

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Composite outcome of Metabolic markers | 6 months
  Fasting blood samples were drawn for the following measurements: serum total cholesterol, HDL-cholesterol (HDL-C), LDL-C, triglycerides, fibrinogen and serum glucose. Serum LDL-C concentration was calculated using the Friedewald equation.
Composite outcome of Anthropometric measurements | 6 months
  BMI was calculated as the ratio of body weight to height2 (kg/m2). Waist circumference was measured with an inelastic tape, the subject in standing position, at the level of the umbilicus. According to the National Cholesterol Education Program (NCEP) Adult Treatment Panel III (ATP III) criteria,abdominal obesity was defined as waist circumference ≥102 cm in men and ≥88 cm in women
Composite outcome of Clinical assessments | 6 months
  Clinical assessment was based on three separate instruments: Psoriasis Area and Severity Index (PASI), Dermatology Life Quality Index (DLQI), and VAS for subjective itch ratings.
  The PASI is used for measuring psoriasis severity. The scale evaluates four areas of the body (head/neck, upper limbs, trunk, and lower limbs) for erythema, scaliness and thickness of psoriatic plaques. The PASI score can range from 0 to 72, with higher scores indicating greater severity.
  The DLQI is a self-rated instrument consisting of ten items related to the ways that skin disease may impact a patient's health-related quality of life (HRQL). Scores are based on six subscales and has a possible range 0 to 30, with 30 corresponding to the worst HRQL.
  Subjective itch ratings were recorded using a computerized VAS, anchored by the terms "no itching" (0 points) and "severe itching" (10 points). Subjects were asked to respond in terms of their itching "at the present time".
Composite outcome of Dietary assessment | 6 months
  Dietary compliance was evaluated by experienced dietitians trained for this project, using a combination of food diaries, personal interviews and a detailed food-frequency questionnaire that included 130 foods and beverages. Information on diet included weekly frequency of consumption and portion size. Average daily intakes were calculated by using food tables and industry estimates of the n-3 naturally-rich margarine. Total dietary n3 PUFAs refers to the intake of ALA in addition to of long-chain EPA and DHA.

CONTACTS AND LOCATIONS:
Locations (1):
- federico II University, Naples, Naples, Italy

REFERENCES:
- [Derived] Guida B, Napoleone A, Trio R, Nastasi A, Balato N, Laccetti R, Cataldi M. Energy-restricted, n-3 polyunsaturated fatty acids-rich diet improves the clinical response to immuno-modulating drugs in obese patients with plaque-type psoriasis: a randomized control clinical trial. Clin Nutr. 2014 Jun;33(3):399-405. doi: 10.1016/j.clnu.2013.09.010. Epub 2013 Sep 28. PMID 24120032